CLINICAL TRIAL: NCT06063694
Title: Prospective Randomized Controlled Trial Comparing Infection Rates and Wound Closure Following Transmetatarsal Amputation With Aid of Electrospun Fiber Matrix
Brief Title: Comparing Wound Complication Following TMA With Aid of Electrospun Fiber Matrix
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Health (Other)
Collaborators: North Park Podiatry (Other)
Responsible Party: Principal Investigator, Trent Brookshier, Principal Investigator, Scripps Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Single application RCT in TMA
Record Dates: First submitted 2023-09-09; First posted 2023-10-02 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Amputation; Wound; Foot; Wound Complication
MeSH Terms: conditions — Foot Injuries

STUDY DESIGN:
Intervention Model Description: Group 1: transmetatarsal amputation without augmentation Group 2: transmetatarsal amputation augmentation with synthetic electrospun fiber matrix
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transmetatarsal amputation with primary closure (No Intervention): Transmetatarsal amputation with primary closure and no application of synthetic electrospun fiber matrix.
- Transmetatarsal amputation with application of synthetic electrospun fiber matrix (Experimental): Transmetatarsal amputation with application of synthetic electrospun fiber matrix
  Interventions: Device: Synthetic electrospun fiber matrix

INTERVENTIONS:
Device: Synthetic electrospun fiber matrix — Electrospun fiber matrices have long been investigated as an innovative construct for use in tissue engineering and regenerative medicine research due to their ability to mimic the structure and scale of native tissue. Clinical studies have demonstrated clinical efficacy in treating both chronic and acute wounds. There is strong evidence to support the application of a synthetic electrospun fiber matrix will generate favorable wound healing and reduce infection rates when used to augment transmetatarsal amputation.
  Other Names: Restrata
  Arms: Transmetatarsal amputation with application of synthetic electrospun fiber matrix

SUMMARY:
Transmetatarsal amputation (TMA) patient populations commonly have poor healing outcomes and a large number of complications. There has been little study on the benefits of augmenting a TMA with a synthetic graft substitute. The long term goal is to push for an application of synthetic graft substitute to reduce infection rates and aid in the healing process. Augmenting a TMA with a synthetic electrospun fiber matrix will demonstrate utilization of the product and other comparators in generating wound healing and infection rate outcomes including rate of infection, wound dehiscence and total healing response. Electrospun fiber matrices have long been investigated as an innovative construct for use in tissue engineering and regenerative medicine research due to their ability to mimic the structure and scale of native tissue. Clinical studies have demonstrated clinical efficacy in treating both chronic and acute wounds. There is strong evidence to support the application of a synthetic electrospun fiber matrix will generate favorable wound healing and reduce infection rates.

DETAILED DESCRIPTION:
Intervention or Exposure

* Transmetatarsal amputation with application of synthetic electrospun fiber matrix
* After surgery, patient will be off-loaded to the surgical site with an off-loading device based on the investigator's decision, e.g., a boot for forefoot and a heel protector for hindfoot. Patients should be instructed on how to care for the surgical site, utilize an off-loading device, and keep the surgical site moist and clean.

Comparison intervention or Exposure

* Transmetatarsal amputation without application of synthetic electrospun fiber matrix
* After surgery, patient will be off-loaded to the surgical site with an off-loading device based on the investigator's decision, e.g., a boot for forefoot and a heel protector for hindfoot. Patients will be instructed on how to care for the surgical site, utilize an off-loading device, and keep the surgical site moist and clean.

Outcomes

* Primary: Infection rate at 1 week postoperative follow-up visit
* Secondary: Wound dehiscence rate and wound healing status at 12 weeks post operatively. Infection rate at 2, 4, and 12 weeks post operatively.
* Patients will have follow-up visits at week 1, 2, 4, and 12. Assessment and imaging of the wound will occur at each visit. Assessment of adverse events, infection, and dehiscence will occur during each visit. Assessment of wound(s) through gross observation and analysis, wound progression, and tissue healing. Gross observation will be utilized to determine the necessity of standard dressing change. Carefully assess the wound(s) for signs of infection, dehiscence, and description of exudate present. Debridement and dressing changes may occur at each weekly visit or as needed. Debride the wound(s) as needed while not disrupting healing tissue. Photographic image will be obtain to document wound appearance. The clinician will inspect the wound bed for signs of infection and healing. Frequency of secondary dressing changes will be dependent upon the volume of exudate produced, type of dressing used and the clinician's decision upon inspection of the wound(s).
* Measurement and imaging of wound(s). If debridement is completed during this visit, then the assessment must be completed after debridement.

Timing of study

* Preop visit for eligibility and randomization
* Surgical visit: TMA with or without application of synthetic electrospun fiber matrix
* 1, 2, 4, and 12 week post-op visits.

Setting of study

* Inpatient at Scripps Mercy Hospital
* Outpatient follow-up Scripps Mercy Podiatry Specialty Clinic or Dr. Brookshier's private clinic North Park Podiatry

Study exit: patient's participation in the study will end after any of the following

* Completion of 12 week follow-up period
* Pathology results from TMA surgery revealing active infection within remaining surgical margins
* Patient withdrawal
* The Investigator may withdraw the patient if he/she determines it is in the patient's best interest
* Patient lost to follow-up
* Amputation of the study limb
* Closure of study
* Patient death

Variables that can be collected: HbA1c, patients that require revascularization prior to TMA due to poor vascular status, age, gender, smoking status

Application of synthetic electrospun fiber matrix (SEFM)

1. Wound Bed Preparation post TMA. Following amputation, prepare the wound bed using standard methods to ensure it is free of devitalized tissue. An initial excision or debridement of the wound is necessary to ensure the wound edges contain viable tissue. Cleanse the wound thoroughly with sterile saline prior to application of SEFM.
2. Preparation of SEFM. Select the appropriate size sheet of SEFM based on the size of the post-amputation defect. Heavily fenestrate with a scalpel or mesh prior to application. SEFM must be fenestrated prior to use in any wound prone to exudate in order to permit effective exudate management. SEFM is packaged in a nested pouch configuration. Peel open the outer foil pouch starting from the chevron sealed edge. The inner pouch is sterile and may be placed on the sterile field. Rinse surgical gloves, if necessary, to remove any glove powder prior to touching the product. SEFM can be cut to the desired shape in a wet or dry state. In order to increase pliability of the product, hydrate in warm, sterile, hypertonic solution (i.e., saline, water, etc.) for a minimum of 1 minute. The matrix should be cut down to fit the size of the wound and applied in full contact with the wound bed.
3. Application of SEFM. Place the SEFM within the surgical defect within the open space. Discard any unused pieces of study product. Management of wound exudate will determine the required dressing. The dressing will be securely in place and dressing determined by provider preference.

Adverse events will be documented. The following adverse events whether or not they are related to a study product/procedure:

* Infection of wound and/or area surrounding wound
* Complete or partial amputation of lower extremity
* Allergic reaction to a study product
* Excessive redness, pain, swelling or blistering of wound

ELIGIBILITY:
Inclusion Criteria:

* Undergoing TMA
* At least 18 years old
* Adequate perfusion demonstrated by either TcPO2 or ankle-brachial index (ABI) or toe-brachia index (TBI) within 60 days prior to enrollment/randomization (Dorsum TcPO2 of study leg(s) ≥40mmHg OR ABI of study leg(s) with results of ≥ 0.7 and ≤ 1.3 OR TBI of study extremity(ies) with results of ≥ 0.5).
* Patient is willing and capable of complying with all protocol requirements.
* Patient or legally authorized representative (LAR) is willing to provide written informed consent prior to any study procedures

Exclusion Criteria:

* Previously enrolled into this study or is currently participating in another prospective drug or device study that has not reached its primary endpoint.
* Patient is pregnant, breast feeding or planning to become pregnant.
* Patient has a known allergy to resorbable suture materials.
* Patient has a life expectancy less than three months as assessed by the investigator.
* Patient has received skin substitutes during the run-in period or within 14 days prior to beginning of run-in period.
* Patient currently undergoing cancer treatment.
* Patient diagnosed with autoimmune connective tissue.
* Patient is taking parenteral corticosteroids or any cytotoxic agents for 7 consecutive days during the run-in period or up to 30 days before the run-in period.
* Chronic oral steroid use is not excluded if dose is <10 mg per day for prednisone.
* Patient unwilling or unable to safely utilize appropriate offloading device to unweight wound(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Infection rate of transmetatarsal amputation site at 1 week postoperative | 1 week post-operatively
  Assessment for signs of infection to transmetatarsal amputation site in both groups at 1 week post-operative follow-up visit.
  * Assess if patient currently on antibiotics
  * Amount of wound exudate (none, scant, small, moderate or large)
  * Type of wound exudate (bloody, serosanguinous, serous, purulent, or foul purulent)
  * Erythema, edema, and/or increased warmth at surgical site
  * Presence of fevers or chills
  * Clinical signs of infection
  * Photographs taken of the surgical site to document appearance
  * Wounds measured in centimeters (length, width, depth)

SECONDARY OUTCOMES:
Infection rate of transmetatarsal amputation site at 2, 4 and 12 weeks postoperative | 2, 4 and 12 weeks postoperatively
  Assessment for signs of infection to transmetatarsal amputation site in both groups at 2, 4 and final 12 weeks post-operative follow-up visit.
  Assessment for signs of infection to transmetatarsal amputation site in both groups at 1 week post-operative follow-up visit.
  * Amount of wound exudate (none, scant, small, moderate or large)
  * Type of wound exudate (bloody, serosanguinous, serous, purulent, or foul purulent)
  * Erythema, edema, and/or increased warmth at surgical site
  * Presence of fevers or chills
  * Clinical signs of infection
  * Wounds measured in centimeters (length, width, depth)
  * Assessments will then be aggregated into yes or no for infection
Wound dehiscence rate of transmetatarsal amputation site at 12 weeks postoperative | 12 weeks postoperatively
  Assess for signs of wound dehiscence in both groups at final 12 weeks postoperative follow-up visit.
  * Photographs taken of the surgical site to document appearance
  * Wounds measured in centimeters (length, width, depth)
  * Assess if surgical edges are intact and well-coapted
  * Assess wound bed condition (necrotic tissue, granulation tissue or epithelialized)
  * If presence of necrotic tissue, assess amount (Not able to visualize; none visible; < 25% of wound covered; 25 to 50% of wound covered; > 50% to 75% of wound covered; 75% to 100% of wound covered)
  * Assessments will then be aggregated into yes or no for wound dehiscence
Wound healing status of transmetatarsal amputation site at 12 weeks postoperative | 12 weeks postoperatively
  Assess final wound healing status in both groups at 12 weeks postoperative follow-up visit.
  * Photographs taken of the surgical site to document appearance
  * Wounds measured in centimeters (length, width, depth)
  * Assess if surgical edges are intact and well-coapted
  * Assess wound bed condition (necrotic tissue, granulation tissue or epithelialized)
  * Assessments will then be aggregated into either fully healed, partially healed, or non-healing.

CONTACTS AND LOCATIONS:
Overall Officials: Trent Brookshier, DPM, Principal Investigator — Scripps Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCallum R, Tagoe M. Transmetatarsal amputation: a case series and review of the literature. J Aging Res. 2012;2012:797218. doi: 10.1155/2012/797218. Epub 2012 Jul 3. PMID 22811912
- [Background] Alexander J, Desai V, Denden S, Alianello N. Assessment of a Novel Augmented Closure Technique for Surgical Wounds Associated with Transmetatarsal Amputation: A Preliminary Study. J Am Podiatr Med Assoc. 2022 Sep-Oct;112(5):20-256. doi: 10.7547/20-256. PMID 36251595
- [Background] MacEwan M, Jeng L, Kovacs T, Sallade E. Clinical Application of Bioresorbable, Synthetic, Electrospun Matrix in Wound Healing. Bioengineering (Basel). 2022 Dec 21;10(1):9. doi: 10.3390/bioengineering10010009. PMID 36671580
- See also: Diabetes and Disability — https://www.ncbi.nlm.nih.gov/books/NBK567983/